CLINICAL TRIAL: NCT06369961
Title: A Retrospective Clinical Study on the Impact of Nutritional Status on the Analgesic Effect of Fentanyl Transdermal Patches in Cancer Pain Patients
Brief Title: Correlation Between the Analgesic Effect of Fentanyl Transdermal Patches and Nutritional Status in Cancer Pain Patients
Status: Completed | Type: Observational
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDFCANCERPAIN20230101
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer Pain; Nutrition Disorders
MeSH Terms: conditions — Cancer Pain; Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Those who used TDF
  Interventions: Drug: transdermal fentanyl

INTERVENTIONS:
Drug: transdermal fentanyl — Adult cancer pain patients switched from oral opioid to TDF

SUMMARY:
The goal of this observational study is to investigate the correlation and quantitative relationship between the analgesic effect of fentanyl transdermal patches in cancer pain patients and their nutritional status.

DETAILED DESCRIPTION:
Cancer-related pain is one of the most common and unbearable symptoms among patients with malignant tumors. Opioids are commonly used to treat moderate or severe cancer pain. Among them, fentanyl is a synthetic opioid with analgesic adjuvant with a 50~100 times higher potency than morphine. Due to its small molecular weight, high lipid solubility, and low irritation to the skin, transdermal fentanyl (TDF) is formulated, which is more convenient for patients with intestinal obstruction, swallowing difficulties, and intolerance to oral opioids. According to some research, the TDF demonstrated good cancer pain control for patients switching from morphine or oral oxycodone preparations, and was well tolerated.

However, a part of patients still go through increased breakthrough pain, sleep disturbances, and even accompanied by anxiety and depression when using TDF. Therefore, early identification of cancer pain patients using TDF at risk of ineffectiveness is an essential step in increasing analgesic effectiveness, and improving quality of life.

Some studies discovered different clinical factors such as age, gender, serum albumin, glomerular filtration rate, kidney disease, body mass index (BMI), total protein, alanine aminotransferases have some influence on fentanyl serum concentration and the dose of TDF. Furthermore, the clinical factors seem to have a greater impact on the effectiveness of TDF than the genetic factors which may affect the liver metabolism of fentanyl. Based on these results, we aim to investigate the correlation and quantitative relationship between the analgesic effect of fentanyl transdermal patches in cancer pain patients and their nutritional status. Our purpose is to help clinicians recognize and increase the analgesic effect of TDF according to the patient's risk level.

ELIGIBILITY:
Inclusion Criteria:

* Cancer pain patients admitted to our hospital;
* Cancer pain patients switched from oral sustained-release strong opioid analgesics to fentanyl transdermal patches during the hospital stay.

Exclusion Criteria:

* Patients who have been switched to fentanyl transdermal patches after titration with an analgesic pump;
* Patients using fentanyl transdermal patches in combination with other oral sustained-release strong opioid analgesics;
* Patients using fentanyl transdermal patches in combination with an analgesic pump;
* Patients who have used fentanyl transdermal patches for less than 3 days;
* Patients with postoperative pain;
* Patients with allergies;
* Patients who are pregnant women;
* Patients with missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient at the oncology hospital
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
11-point numeric rating scale (NRS) after TDF treatment | in 1 week
  Ineffectiveness defined as pain with a NRS of 4 or higher.
the occasions that breakthrough pain attacks per day after TDF treatment | in 1 week
  Ineffectiveness defined as the breakthrough pain attacks more than 3 occasions per day
The dose adjustment of TDF | in 1 week
  Ineffectiveness defined as the dosage of TDF increased
The kinds of other analgesics combined with TDF | in 1 week
  Ineffectiveness defined as more than one kind of analgesics were combined with TDF

SECONDARY OUTCOMES:
Adverse effects | in 1 week
  Nausea, vomiting, dizziness, rash, constipation, urinary retention, respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: Chao Li, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chao Li, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Minello C, George B, Allano G, Maindet C, Burnod A, Lemaire A. Assessing cancer pain-the first step toward improving patients' quality of life. Support Care Cancer. 2019 Aug;27(8):3095-3104. doi: 10.1007/s00520-019-04825-x. Epub 2019 May 11. PMID 31076899
- [Result] Barratt DT, Bandak B, Klepstad P, Dale O, Kaasa S, Christrup LL, Tuke J, Somogyi AA. Genetic, pathological and physiological determinants of transdermal fentanyl pharmacokinetics in 620 cancer patients of the EPOS study. Pharmacogenet Genomics. 2014 Apr;24(4):185-94. doi: 10.1097/FPC.0000000000000032. PMID 24469018
- [Result] Moryl N, Bokhari A, Griffo Y, Hadler R, Koranteng L, Filkins A, Zheng T, Horn SD, Inturrisi CE. Does transdermal fentanyl work in patients with low BMI? Patient-reported outcomes of pain and percent pain relief in cancer patients on transdermal fentanyl. Cancer Med. 2019 Dec;8(18):7516-7522. doi: 10.1002/cam4.2479. Epub 2019 Sep 30. PMID 31568684
- [Derived] Chen Y, Han S, Hu X, Ma X, Qiu Y, Tang Y, Wang X, Li L, Li C, Chen W. High BMI predicts poor cancer pain relief when rotating from oral opioids to transdermal Fentanyl: a two-center retrospective study. Pharmacol Rep. 2025 Jun;77(3):789-799. doi: 10.1007/s43440-025-00723-8. Epub 2025 Apr 11. PMID 40214947